CLINICAL TRIAL: NCT01397448
Title: Prevention of Recurrent Gastric or Duodenal Ulcers Caused by Low-dose Aspirin With Rabeprazole (E3810) Treatment. - A Multicenter, Randomized, Parallel-group, Double-blind Comparative Trial-
Brief Title: Prevention of Recurrent Gastric or Duodenal Ulcers Caused by Low-dose Aspirin With Rabeprazole (E3810) Treatment (Planetarium Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: E3810-J081-308
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-10

CONDITIONS: Gastric or Duodenal Ulcers Caused by Low-dose Aspirin
Keywords: Rabeprazole; proton pump inhibitor; Acetylsalicylic Acid; Aspirin; Gastric Ulcer; Duodenal Ulcer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Rabeprazole; geranylgeranylacetone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- E3810 5 mg (Experimental)
  Interventions: Drug: E3810
- E3810 10 mg (Experimental)
  Interventions: Drug: E3810
- Teprenone 150 mg (Active Comparator)
  Interventions: Drug: Teprenone

INTERVENTIONS:
Drug: E3810 — E3810 5 mg/day Group: Orally administered E3810 5 mg tablets and E3810 10 mg placebo tablets once daily after breakfast; and orally administered Teprenone 50 mg placebo capsules three times daily after each meal.
  Arms: E3810 5 mg
Drug: E3810 — E3810 10 mg Group: Orally administered E3810 5 mg placebo tablets and 10 mg tablets once daily after breakfast; and orally administered Teprenone 50 mg placebo capsules three times daily after each meal.
  Arms: E3810 10 mg
Drug: Teprenone — Teprenone 150 mg/day Group: Orally administered E3810 5 mg placebo tablets and 10 mg placebo tablets once daily after breakfast; and orally administered Teprenone 50 mg capsules three times daily after each meal.
  Arms: Teprenone 150 mg

SUMMARY:
The primary objective of this study to evaluate the effect of preventing recurrence of gastric or duodenal ulcers by administering E3810 5 mg or 10 mg tablets once daily or Teprenone 150 mg/day (50 mg three times daily) as a control to patients receiving low-dose aspirin and thereby examine the superiority of E3810 over Teprenone.

ELIGIBILITY:
Inclusion Criteria

* Require long-term administration of low-dose aspirin (81 mg/day or 100 mg/day)
* Confirmed to have a history of gastric or duodenal ulcer

Exclusion Criteria

-Confirmed to have acute gastro duodenal mucosal lesions, gastric or duodenal ulcer, or upper gastrointestinal (esophagus, stomach, duodenum) bleeding Confirmed to have reflux esophagitis or long segment Barrett's esophagus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sugisaki, Study Director — Japan/Asia Clinical Research Product Creation Unit
Locations (49):
- Japan (49):
  - Kasugai, Aichi-ken
  - Nagoya, Aichi-ken
  - Ichikawa, Chiba
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Gifu, Gifu
  - Maebashi, Gunma
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Itami, Hyōgo
  - Kobe, Hyōgo
  - Hitachi, Ibaraki
  - Fujisawa, Kanagawa
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Hitoyoshi, Kumamoto
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Ebino, Miyazaki
  - Miyazaki, Miyazaki
  - Chikuma, Nagano
  - Matsumoto, Nagano
  - Nagano, Nagano
  - Suzaka, Nagano
  - Nagasaki, Nagasaki
  - Beppu, Oita Prefecture
  - Ōita, Oita Prefecture
  - Yufu, Oita Prefecture
  - Daitō, Osaka
  - Hirakata, Osaka
  - Matsubara, Osaka
  - Osaka, Osaka
  - Takatsuki, Osaka
  - Yao, Osaka
  - Karatsu, Saga-ken
  - Saga, Saga-ken
  - Ureshino, Saga-ken
  - Izumo, Shimane
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Ohtawara, Tochigi
  - Mitaka, Tokyo
  - Setagaya City, Tokyo
  - Shinjuku, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Rabeprazole 5 mg: Orally administered E3810 (Rabeprazole) 5mg tablet and E3810 10mg placebo tablet once daily after breakfast; and orally administered Teprenone 50mg placebo capsule three times daily after each meal.
- Rabeprazole 10 mg: Orally administered E3810 (Rabeprazole) 5mg placebo tablet and 10mg tablet once daily after breakfast; and orally administered Teprenone 50mg placebo capsule three times daily after each meal.
- Teprenone 150 mg: Orally administered E3810 (Rabeprazole) 5mg placebo tablet and 10mg placebo tablet once daily after breakfast; and orally administered Teprenone 50mg capsule three times daily after each meal.
Period: Overall Study
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg | Teprenone 150 mg
Started | 156 | 157 (158 participants were randomized but 1 participant was not treated with drug.) | 158
Completed | 138 | 142 | 140
Not Completed | 18 | 15 | 18
Not completed — Adverse Event | 4 | 4 | 6
Not completed — Withdrawal by Subject | 4 | 4 | 3
Not completed — Lack of Efficacy | 2 | 0 | 5
Not completed — Other | 8 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg | Teprenone 150 mg | Total
Number analyzed (Participants) | 156 | 157 | 158 | 471
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (8.9) | 70.1 (9.6) | 69.4 (7.9) | 69.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 41 | 112
  Male | 121 | 121 | 117 | 359
Antiplatelet Drug or Anticoagulant Drug [Number; unit: Participants]
  Yes | 30 | 34 | 35 | 99
  No | 126 | 123 | 123 | 372
Daily Dose of Low-Dose Aspirin [Number; unit: Participants]
  81 mg | 12 | 14 | 16 | 42
  100 mg | 144 | 143 | 142 | 429
Diagnostic Test of H.pylori. (IgG Antibody) [Number; unit: Participants]
  Positive | 72 | 67 | 77 | 216
  Negative | 84 | 90 | 81 | 255
Primary Disease [Number; unit: Participants] — Percutaneous Transluminal Coronary Angioplasty is represented as PTCA.
  Participants
    Angina Pectoris (Yes) | 68 | 63 | 66 | 197
    Angina Pectoris (No) | 88 | 94 | 92 | 274
    Myocardial Infarction (Yes) | 27 | 31 | 33 | 91
    Myocardial Infarction (No) | 129 | 126 | 125 | 380
    Ischemic Cerebrovascular Disease (Yes) | 79 | 77 | 78 | 234
    Ischemic Cerebrovascular Disease (No) | 77 | 80 | 80 | 237
    Coronary Arterial Bypass Grafting or PTCA (Yes) | 52 | 51 | 48 | 151
    Coronary Arterial Bypass Grafting or PTCA (No) | 104 | 106 | 110 | 320
    Other (Yes) | 6 | 10 | 9 | 25
    Other (No) | 150 | 147 | 149 | 446

OUTCOME MEASURES:

1. Secondary Outcome: Cumulative Incidence of Bleeding Ulcers
Time Frame: 24 weeks
Population: Defined as all randomized participants who received at least one dose of the study drug and showed no ulcers at baseline, and from whom the results of at least one endoscopic assessment was available.
Measure: Number (95% Confidence Interval); unit: Events/100 participants/24 weeks
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg | Teprenone 150 mg
Number analyzed (Participants) | 150 | 151 | 151
Events/100 participants/24 weeks | 0 [0 to 0] | 0 [0 to 0] | 4.6 [2.24 to 9.48]

2. Primary Outcome: Cumulative Recurrent Rates of Gastric or Duodenal Ulcers
Description: Mucosal injuries with a white coat measuring 3 mm in diameter will be diagnosed as ulcers. When ulcer is confirmed by endoscopic examination during the trial, it will be regarded as recurrence of ulcer and the trial will be discontinued for the patient involved.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events/100 participants/24 weeks
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg | Teprenone 150 mg
Number analyzed (Participants) | 150 | 151 | 151
Events/100 participants/24 weeks | 2.8 [1.04 to 7.17] | 1.4 [0.35 to 5.51] | 21.7 [15.84 to 29.27]
Statistical Analysis 1: Comparison: Rabeprazole 5 mg vs Teprenone 150 mg; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.11, 95% CI 2-sided [0.04 to 0.31]
Statistical Analysis 2: Comparison: Rabeprazole 10 mg vs Teprenone 150 mg; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.05, 95% CI 2-sided [0.01 to 0.23]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg | Teprenone 150 mg
Serious Adverse Events (participants affected / at risk) | 10/156 | 6/157 | 10/158
Other Adverse Events (participants affected / at risk) | 48/156 | 46/157 | 41/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 5 mg (N=156) | Rabeprazole 10 mg (N=157) | Teprenone 150 mg (N=158)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 5 mg (N=156) | Rabeprazole 10 mg (N=157) | Teprenone 150 mg (N=158)
Constipation (Gastrointestinal disorders) | 1 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 6 | 2
Nasopharyngitis (Infections and infestations) | 25 | 22 | 25
Pharyngitis (Infections and infestations) | 6 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 6 | 1
Hypertension (Vascular disorders) | 0 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.